CLINICAL TRIAL: NCT06238310
Title: Comparison of Two Different External Clearance Markers for Measuring Glomerular Filtration Rate (GFR) - Mannitol and Iohexol, in Patients Treated in the Intensive Care Units and in Outpatients With Chronic Kidney Disease.
Brief Title: Comparison of Two Different External Clearance Markers - Mannitol and Iohexol for Measuring Glomerular Filtration Rate
Acronym: GFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katalin Kiss (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Katalin Kiss, consultant anesthesiologist, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mannitol GFR
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury; Chronic Kidney Insufficiency
Keywords: Glomerular Filtration Rate
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients in the intensive care unit and outpatients with acute or chronic kidney insufficiency (Experimental): Measuring glomerular filtration rate (GFR) with two different marker and the same measuring protocol.
  Interventions: Diagnostic Test: Comparison of two external marker substance for measuring glomerular filtration rate

INTERVENTIONS:
Diagnostic Test: Comparison of two external marker substance for measuring glomerular filtration rate — Two external marker substance compares for measuring GFR.

SUMMARY:
GFR is the best parameter of the real kidney function. Measurements, however are time-consuming and have limited capacity.

Patients treated in the intensive care units often have more than one organ-insufficiency and acute kidney injury (AKI) has an incidence of up to 70 %. GFR changes dynamically and this is one of the reasons why GFR-measurements have limited indications on the ICU. Retention of medicines or their active metabolites, however can lead to side effects, toxicity and or prolonged ICU-stay. Moreover, patients with allergy to actually standard marker, contrast material iohexol, or gravid patients are not candidate for measuring GFR with iohexol.

In this prospective clinical trial two exogen marker substances will be compared, mannitol as a new marker and iohexol as a standard marker for measuring glomerular filtration rate (GFR). Patients in the intensive care units (ICU) and an outpatient group with stable chronic kidney disease (CKD) are included.

The main question is, how reliable mannitol-GFR is compared to iohexol-GFR in a wide range of kidney insufficiency.

GFR measurements are performed with a bolus injection technique. Patients get mannitol and iohexol bolus at time zero and blood samples are taken three times according to local protocols for iohexol clearance measurements.

DETAILED DESCRIPTION:
Written inform consent from the patients or their relatives if they can not communicate.

Inclusion criteria:

Patients with acute or acute on chronic kidney failure (AKI, CKD), who are treated in the intensive care units because of any kind of organ insufficiency are enrolled. Stabil circulatory parameters needed with or without vasoactive drugs. Continuous intravenous administration of fluids and drugs without significant changes during the study period.

Exclusion criteria:

Unstable circulation and need for fluid resuscitation. Known extracellular volume expansion as ascites or peripheral edema. Intravenous paracetamol administration between or during the measurement period. Measurement with iohexol as contrast material during the previous days. Missing inform consent. Allergy to contrast material.

Sample taking: at time zero and three times after the bolus injection. Timing is scheduled according to the local protocol for iohexol-GFR calculation. Samples are coded and can not identified when results are published.

Outcome measures: Is mannitol clearance a reliable method for measuring GFR compared to iohexol-clearance? Comparing the two methods with Bland-Altman plots and statistical calculation for accuracy P30 and P20.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or acute on chronic kidney failure (AKI, CKD) on intensive care units because of any kind of organ insufficiency.
* Stabile circulatory parameters.
* CKD-patients in outpatient group

Exclusion Criteria:

* unstable circulation with need for fluid resuscitation.
* known extracellular volume expansion as ascites or peripheral edema.
* Intravenous paracetamol administration between or during the measurement period.
* measurement with iohexol during the previous days.
* missing inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Measuring GFR with two different external markers, mannitol as new and iohexol as standard marker | 12 weeks
  Bland-Altman statistic is used for result comparison and Accuracy, P30 and P20 is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Bragadottir, MD, PhD, Study Director — Department of Cardiothoracic Surgery, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- SahlgrenskaUH, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhont E, Windels C, Snauwaert E, Van Der Heggen T, de Jaeger A, Dhondt L, Delanghe J, Croubels S, Walle JV, De Paepe P, De Cock PA. Reliability of glomerular filtration rate estimating formulas compared to iohexol plasma clearance in critically ill children. Eur J Pediatr. 2022 Nov;181(11):3851-3866. doi: 10.1007/s00431-022-04570-0. Epub 2022 Sep 2. PMID 36053381
- [Result] Kiss K, Molnar M, Sondergaard S, Molnar G, Ricksten SE. Mannitol clearance for the determination of glomerular filtration rate-a validation against clearance of 51 Cr-EDTA. Clin Physiol Funct Imaging. 2018 Jan;38(1):10-16. doi: 10.1111/cpf.12374. Epub 2016 Jun 3. PMID 27256921